CLINICAL TRIAL: NCT06634147
Title: Prevention of Functional and Cognitive Impairment Through a Multicomponent Exercise Program in Hospitalized Older Adults (Geriatrics and Internal Medicine): a Randomized Clinical Trial. Multicenter Study (HUN, CHU-T, ULSBM, and HNSM)
Brief Title: Prevention of Functional and Cognitive Impairment Through a Multicomponent Exercise Program in Hospitalized Older Adults
Acronym: PREDISC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREDISC
Record Dates: First submitted 2024-09-03; First posted 2024-10-09 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Clinical Deterioration
Keywords: hospital acquired disability; exercise; function; cognition
MeSH Terms: conditions — Clinical Deterioration; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Multicenter Randomized Clinical Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No exercise during hospitalization
- Intervention group (Experimental): Exercise during hospitalization
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Multicomponent individualized exercise intervention As mentioned earlier, patients in the control group (G0) will receive the usual care currently provided to other patients, which includes a referral to physical therapy if needed.
  The intervention for the multicomponent physical exercise intervention group (G1) will consist of a multicomponent physical training program that includes progressive and supervised aerobic endurance, strength, and balance training lasting 4-7 days during their hospitalization. This will be supervised by the research team from the Geriatrics Unit. Additionally, after hospital discharge, they will receive individualized guidelines to engage in multicomponent physical exercise for 3 months, along with individualized recommendations from the Nutrition and Dietetics Service of HUN.
  The multicomponent physical training program will consist of chair squat exercises. The main part of the training will utilize machines for strength training for the lower extremit
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to determine whether a multicomponent exercise program improves functional capacity and cognitive status in hospitalized elderly patients aged 75 and older. Additionally, the study aims to assess the impact of this program on medication use, quality of life, and overall health outcomes. Key questions include whether the program enhances functional and cognitive capacities and which subgroups benefit most, such as frail patients or those with cognitive impairment.

Participants will engage in a structured exercise program that includes strength training, balance exercises, and walking, all designed to improve mobility and reduce fall risk. They will attend supervised sessions several times a week, allowing for individualized attention and adjustments based on their abilities and health status.

Throughout the study, changes in functional capacity will be monitored using standardized assessments that measure mobility, strength, and overall physical functioning. Cognitive assessments will evaluate any changes in cognitive status during the intervention and follow-up periods post-discharge. Participants will provide information on medication usage to analyze whether the exercise program can reduce the need for medications or help manage common polypharmacy issues.

Surveys and interviews will assess participants' quality of life, including physical, emotional, and social well-being, before and after the intervention. Follow-up assessments will track progress and outcomes, ensuring long-term benefits of the exercise program are documented.

The study will include a diverse sample from multiple centers, focusing on individuals aged over 75 who are hospitalized in Geriatrics and Internal Medicine services across participating centers (HUN, CHU-T, ULSBM, and HNSM). Exclusion criteria will ensure safety, excluding those with terminal illnesses or significant contraindications for exercise.

This clinical trial aims to recruit 296 patients, providing valuable insights into the benefits of physical activity for elderly patients during hospitalization and informing future care practices.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if a multicomponent exercise program improves functional capacity and cognitive status in hospitalized elderly patients aged 75 and older. Additionally, the study aims to assess the impact of this program on medication use, quality of life, and the overall health outcomes of these patients. The main questions it aims to answer are:

1. **Does the multicomponent exercise program enhance functional capacity in hospitalized elderly patients?**
2. **Which subgroups of patients benefit the most from the intervention (e.g., frail patients, those with cognitive impairment, or malnutrition)?**
3. **Does participation in the exercise program lead to a reduction in the consumption of medications and instances of iatrogenic complications?**
4. **How does the exercise program affect the quality of life and sleep quality of the participants?**
5. **What are the long-term effects of the exercise intervention on muscle mass, balance, and walking speed?**
6. **Are there measurable changes at the omics level (genomic, proteomic, metabolomic) due to the exercise intervention?**

Researchers will compare the multicomponent exercise program to standard care to see if the exercise program leads to significant improvements in functional and cognitive outcomes. This comparison will help determine the effectiveness of the exercise intervention in enhancing the overall well-being of elderly patients during their hospital stay.

**Participants will:**

* Engage in a structured multicomponent exercise program designed specifically for elderly patients. This program will include activities focused on strength training, balance exercises, and walking to improve mobility and reduce the risk of falls. The exercises will be tailored to the individual capabilities of each participant, ensuring safety and effectiveness.
* Attend supervised exercise sessions several times a week, allowing for individualized attention and adjustments based on each participant's abilities and health status. These sessions will be conducted by trained physical therapists who specialize in geriatric care.
* Be monitored for changes in functional capacity using standardized assessments, which will measure improvements in mobility, strength, and overall physical functioning. Assessments will include tools such as the Timed Up and Go Test (TUG), the Berg Balance Scale, and the 6-Minute Walk Test.
* Undergo cognitive assessments to evaluate any changes in cognitive status throughout the intervention and during follow-up periods after discharge. Cognitive evaluations will include tests like the Mini-Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA).
* Provide information on their medication usage to analyze whether the exercise program can reduce the need for medications or help manage polypharmacy issues commonly faced by elderly patients. This will include a detailed review of current medications and any changes made during the study.
* Participate in surveys and interviews to assess their quality of life, including physical, emotional, and social well-being, before and after the intervention. Quality of life will be measured using validated tools such as the Short Form Health Survey (SF-36) and the EuroQol-5D (EQ-5D).
* Attend follow-up assessments at designated intervals to track their progress and outcomes, ensuring that any long-term benefits of the exercise program are recognized and documented. Follow-ups will occur at 1 month, 3 months, and 6 months post-discharge.

The study will include a diverse sample of participants from multiple centers, ensuring a robust analysis of the intervention's effects across different populations. Inclusion criteria will focus on individuals aged over 75 years who are hospitalized in Geriatrics and Internal Medicine services across participating centers (HUN, CHU-T, ULSBM, and HNSM). Participants must be capable of communication and ambulation, either independently or with assistance.

Exclusion criteria will ensure the safety and appropriateness of the intervention. Individuals who explicitly refuse to participate or cannot provide informed consent will be excluded. Additionally, those with a life expectancy of less than three months, terminal illnesses, or significant medical contraindications for exercise will not be eligible. Participants with moderate to severe neurocognitive disorders or disabilities that severely limit mobility will also be excluded to maintain the integrity of the intervention.

**Sample Size and Recruitment:** This clinical trial aims to recruit a total of 296 patients across the four participating centers. Recruitment will be conducted through hospital admissions, with potential participants identified by medical staff and referred to the research team. Informed consent will be obtained from all participants or their legal representatives prior to enrollment.

**Data Collection and Analysis:** Data will be collected at baseline, during the intervention, and at follow-up assessments. This will include demographic information, clinical history, baseline functional and cognitive assessments, and post-intervention evaluations. Statistical analyses will be performed to compare outcomes between the intervention and control groups, using appropriate methods to account for potential confounding factors.

**Ethical Considerations:** This study will adhere to ethical guidelines for research involving human subjects. The protocol will be reviewed and approved by the Institutional Review Board (IRB) at each participating center. Informed consent will be obtained from all participants, ensuring they understand the study's purpose, procedures, risks, and benefits.

**Expected Outcomes:** The findings of this study may provide valuable insights into the benefits of physical activity for elderly patients during hospitalization. By examining the outcomes related to functional capacity, cognitive status, medication use, and quality of life, the study seeks to inform future guidelines and practices for improving the care and rehabilitation of older adults in hospital settings. Additionally, the research may contribute to the understanding of how exercise interventions can positively impact health at the molecular level, potentially leading to new therapeutic approaches for managing health in elderly populations.

Ultimately, the results of this clinical trial could have significant implications for enhancing the quality of care for hospitalized elderly patients, reducing the burden of functional decline, and improving overall health outcomes in this vulnerable population. By demonstrating the effectiveness of a multicomponent exercise program, the study could advocate for the integration of such programs into standard hospital care for older adults, promoting healthier aging and better recovery from acute medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 75 years, admitted to the acute care unit for medical conditions.

Exclusion Criteria:

* Explicit refusal expressed verbally or refusal to sign the informed consent by the patient/main caregiver/legal guardian or inability to obtain it.
* Life expectancy of less than 3 months or terminal oncological or non-oncological disease.
* Inability to follow up.
* Inability to participate in a multicomponent exercise program.
* Medical contraindication to exercise.
* Major neurocognitive disorder at moderate to severe stage (GDS - Fast Reisberg 5-7).
* Moderate to severe disability (measured by the Barthel Index (BI <60)).
* Expected hospital stay of less than 6 days.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional status | Through study completion, an average of 3 months
  Short Performance Physical Battery (SPPB)

SECONDARY OUTCOMES:
Barthel Index | Through study completion, an average of 3 months
  Basic activities of daily living
Mini-Mental State Examination (MMSE) | Through study completion, an average of 3 months
  Cognition
Gait Speed. | Through study completion, an average of 3 months
  Gait Speed (m/sec)
Trail Making Test A | Through study completion, an average of 3 months
  Complex attention
GDS Yesavage | Through study completion, an average of 3 months
  Depression
EuroQol-5D-3L | Through study completion, an average of 3 months
  Quality of life
Number of medications | Through study completion, an average of 3 months
  Number of medications before and after de intervention
Falls | Through study completion, an average of 3 months
  Number of falls during the study
Mortality | Through study completion, an average of 3 months
  Mortality during the study
Hospital Readmissions | Through study completion, an average of 3 months
  Number of hospital readmissions
Hand Grip | Through study completion, an average of 3 months
  Maximum isometric strength
Length of stay | After hospitalization
  Average length of hospital stay
SATED scale | Through study completion, an average of 3 months
  Changes in sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: NICOLAS Martinez-Velilla, PhD, Principal Investigator — Navarrabiomed-Fundación Miguel Servet-Hospital de Navarra
Locations (2):
- Spain (2):
  - Hospital Universitario de Navarra - Navarrabiomed, Pamplona, Navarre
  - Hospital Universitario de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Yes
Clinical, demographic, outcomes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years after the completion of the study
Access Criteria: Data Sharing Agreement: Establish a formal data sharing agreement outlining the terms of use, responsibilities, and conditions for accessing the IPD. This can help protect participant confidentiality and ensure compliance with ethical standards.
  Secure Data Repository: Utilize a secure data repository or platform (e.g., Open Science Framework, Dryad) where researchers can access the IPD. This platform should have robust security measures to protect sensitive data.
  Anonymization Procedures: Implement procedures to anonymize the data before sharing. This may include removing identifiable information and aggregating data to prevent re-identification of participants.
  Access Criteria: Define clear criteria for who can access the IPD. This could include stipulations that only qualified researchers with relevant expertise can apply for access.

REFERENCES:
- [Background] Martinez-Velilla N, Abizanda P, Gomez-Pavon J, Zambom-Ferraresi F, Saez de Asteasu ML, Fiatarone Singh M, Izquierdo M. Effect of an Exercise Intervention on Functional Decline in Very Old Patients During Acute Hospitalizations: Results of a Multicenter, Randomized Clinical Trial. JAMA Intern Med. 2022 Mar 1;182(3):345-347. doi: 10.1001/jamainternmed.2021.7654. PMID 35040873
- [Background] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Saez de Asteasu ML, Lucia A, Galbete A, Garcia-Baztan A, Alonso-Renedo J, Gonzalez-Glaria B, Gonzalo-Lazaro M, Apezteguia Iraizoz I, Gutierrez-Valencia M, Rodriguez-Manas L, Izquierdo M. Effect of Exercise Intervention on Functional Decline in Very Elderly Patients During Acute Hospitalization: A Randomized Clinical Trial. JAMA Intern Med. 2019 Jan 1;179(1):28-36. doi: 10.1001/jamainternmed.2018.4869. PMID 30419096
- [Derived] Martinez-Velilla N, Santos Silva R, Rodriguez PA, Xandri JM, Pais A, Rodriguez EU, Abellan van Kan G, Peyrusque E, Izco-Cubero M, Gonzalez de la Riva MF, Belo R, Zambom-Ferraresi F, Beistegui IE, Chenhuichen C, Galbete A, Gomes AI, Heras E, Zambom-Ferraresi F. Prevention of functional and cognitive impairment through a multicomponent exercise program during and after hospitalization of older adults (PREDISC): Study protocol for a multicenter randomized clinical trial. PLoS One. 2025 Sep 25;20(9):e0332391. doi: 10.1371/journal.pone.0332391. eCollection 2025. PMID 40997056